CLINICAL TRIAL: NCT00764530
Title: Keramos Ceramic/Ceramic Total Hip System
Brief Title: Cementless Alumina-Alumina Total Hip and Hybrid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Encore Medical, L.P. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Study 100
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis; Post-traumatic Arthritis; Avascular Necrosis
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Osteonecrosis | interventions — Reference Standards

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational (Experimental): CeramTec Acetabular Alumina Insert and CeramTec Alumina head used with Foundation Porous Coated Acetabular Shell.
  Interventions: Device: Alumina/Alumina
- Control Device (Active Comparator): Foundation Porous Coated Acetabular Shell with Polyethylene Insert with the CeramTec Alumina head.
  Interventions: Device: Standard

INTERVENTIONS:
Device: Alumina/Alumina — CeramTec Acetabular Alumina Insert and CeramTec Alumina head used with Foundation Porous Coated Acetabular Shell
  Arms: Investigational
Device: Standard — Foundation Porous Coated Acetabular Shell with Polyethylene Insert with the CeramTec Alumina head
  Arms: Control Device

SUMMARY:
Evaluate the safety and efficacy of the CeramTec Acetabular Alumina Insert and CeramTec Alumina head when used with the Foundation Porous Coated Acetabular Shell and an Encore hip stem.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inflammatory tissue disorders (e.g. rheumatoid arthritis, lupus, etc), osteoarthritis, post-traumatic arthritis or secondary arthritis, or avascular necrosis.
* Less than 70 on preoperative HHS score
* Primary total hip replacement
* Patient is likely to be available for evaluation for the duration of the study.

Exclusion Criteria:

* Patients with physical conditions that would eliminate adequate implant support or prevent the use of an appropriately sized implant (e.g., tumor)
* Previous surgery that has adversely affected bone stock (such as some hip pinning or some osteotomies) or prior total hip replacement.
* Insufficient quality or quantity of bone resulting from conditions such as:

  * Cancer, where radiation has destroyed the available bonestock
  * Congenital dislocation
  * Metabolic bone disease of the upper femur or pelvis
  * Femoral osteotomy revision
  * Girdlestone revision
  * Active infection of the hip joint
  * Old or remote infection
  * Other conditions that lead to inadequate skeletal fixation
* Neurological conditions that might hinder patient's ability to follow study procedures, e.g., to restrict physical activities (e.g., Severe Parkinson's, CVA on affected side)
* Patient's mental condition that may interfere with his ability to give an informed consent or willingness to fulfill the required follow-up of the study

  * Mental illness
  * Senility
  * Drug Abuse
  * Alcoholism
* Conditions that place excessive demands on the implant

  * Charcot's joints
  * Muscle deficiencies
  * Multiple joint disabilities
  * Refusal to modify postoperative physical activities
  * Skeletal immaturity
  * Obesity (50% over recorded body weight mass index)
* Greater than or equal to 70 on preoperative HHS score

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2003-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Alumina/Alumina articulation will perform as well as the alumina/polyethylene. | 5 year

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mark Newman, Inc., Newport Beach, California
  - Charleston Orthopaedic Assoc., Charleston, South Carolina
  - Advanced Orthopaedic Centers, Richmond, Virginia

REFERENCES:
- See also: Sponsor company home page — http://www.djosurgical.com